CLINICAL TRIAL: NCT00731445
Title: Phase I/II Dose Escalation, Pharmacokinetic, Safety, and Efficacy Study of Oral Z-208 in Patients With Advanced Hepatocellular Carcinoma
Brief Title: Phase I/II Study of Z-208 in Advanced Hepatocellular Carcinoma (HCC)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zeria Pharmaceutical (Industry)
Responsible Party: Zeria Pharmaceutical Co., Ltd
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07010101
Record Dates: First submitted 2008-08-08; First posted 2008-08-11 (Estimated); Last update posted 2012-07-03 (Estimated); Status verified 2012-06

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: Z-208

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Z-208 — Oral pills taken daily; 8mg, 12mg, 16mg, 4mg

SUMMARY:
This phase I/II is studying the side effect and best dose of Z-208 for patients with advanced hepatocellular carcinoma

DETAILED DESCRIPTION:
This is an open-label, dose-escalation study PhaseI Treatments repeats for 28 days for 1 course in the unacceptable toxicity

Cohort of 3 patients receive escalating doses of Z-208 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 1 of 3 patients experience dose-limiting toxicity.

PhaseII Treatments repeats for 28 days for 6 courses until absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion criteria:

* Histologically or cytologically confirmed hepatocellular carcinoma
* At least one measurable site of disease according to RECIST criteria that has not been irradiated.
* Child-Pugh classification A & B
* ECOG performance status of 0-1
* Life expectancy is more than 90 days
* Adequate organ function as defined by the following criteria, Hemoglobin ≥ 8.0 g/dL WBC ≥ 3,000/mm^3 <12,000/mm^3 Absolute neutrophil count ≥ 1,500/mm^3 Platelet count ≥ 50,000/mm^3 AST and ALT ≤ 5 times upper limit of normal (ULN) Albumin ≥ 2.8 g/dL Bilirubin ≤ 2.0 mg/dL Creatinine ≤ 1.5 times ULN
* Must provide written informed consent prior to the implementation of any study assessment or procedures

Exclusion criteria

* Patients received treatment with any of the following within the specified timeframe;Any surgical procedure, radiofrequency ablation, intraarterial chemotherapy within 30 days prior to signing the ICF, any treatment with transfusion, albumin preparation, G-CSF within 15 days prior to signing the ICF
* CNS involvement must have completed appropriate treatment
* Prior deep vein thrombosis
* Has ascites, pleural effusions or pericardial fluid refractory
* Active clinically serious infection excluding chronic hepatitis
* Any history of deep vein thrombosis, pulmonary embolism, myocardial infraction, cerebrovascular accident
* Allergy or hypersensitivity to Vitamin A
* Women who are pregnant or breast feeding

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2008-07; Primary Completion 2012-01 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Phase I: Determine the maximum tolerated dose (MTD) of Z-208 in patients with advanced hepatocellular carcinoma | 28 days
Phase II : Assess the objective tumor response rate in patients according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria | 28 days for 6 courses

SECONDARY OUTCOMES:
Phase I : Assess the objective tumor response rate in patients according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria | 28 days for 6 courses
Phase I : Determine the pharmacokinetics of this drug in these patients | 28 days for 6 courses
Phase I : Determine the adverse effects profile of this drug in these patients | 28 days for 6 courses
Phase II: Determine the PFS | 28 days for 6 courses

CONTACTS AND LOCATIONS:
Overall Officials: Masao Omata, PhD, MD, Study Chair — Tokyo University
Locations (1):
- The University of Tokyo Hospital, Tokyo, Japan